CLINICAL TRIAL: NCT04490590
Title: A Clinical Trial of Chidamide Combined With Etoposide in Relapsed or Refractory NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, The director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20180814
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: NK/T-Cell Lymphoma
Keywords: Chidamide combined with Etoposide; ORR; CR; PR; TTR; DOR; PFS
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Chidamide+ Etoposide capsule (Experimental): Chidamide: 30mg, twice a week(BIW), PO.
  Etoposide capsule:50mg, quaque die （QD）, PO, d1-10，21days for one cycle. Patients receive the other treatment of chidamide and etoposide capsule, and those who have achieved PD(progressive disease) will give the other treatment.
  Interventions: Drug: Chidamide+ Etoposide

INTERVENTIONS:
Drug: Chidamide+ Etoposide — Patients will receive the treatment of and chidamide and etoposide capsule, and those who have achieved CR（complete response）or PR（partial response）or SD(stable disease)will continue the treatment.

SUMMARY:
To observe the safety, tolerability and clinical effects of Chidamide Combined With Etoposide in Relapsed or Refractory NK/T-cell Lymphoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, one-arm, single center clinical trial, aimed to evaluate the safety, tolerability, and efficacy of Chidamide Combined With Etoposide in Relapsed or Refractory NK/T-cell Lymphoma. A total of 30 patients are planned to be enrolled into the study. Patients with diagnosis of Relapsed or Refractory NK/T-cell Lymphoma will be treated with Chidamide plus Etoposide capsules. The primary end points are objective responder rate (ORR) and a time to response(TTR) and response duration (DOR) and progression free survival(PFS) and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1.age:10-65 years;Eastern Cooperative Oncology Group (ECOG)score≤2;expected survival≥3 months 2 patients with NK/T Cell Lymphoma diagnosed by immuno-histochemistry (IHC) or fluorescence in situ hybridization (FISH); 3.Refractory or relapse after at least 2 regimen 4.Once the patient received radiotherapy, need to be more than 3 months away from this treatment, and it is a non-primary recurrence; 5.No chemotherapy contraindications: hemoglobin ≥ 100g / L, absolute neutrophil count ≥ 1.5 × 109 / L, platelets ≥ 80 × 109 / L, ALT, AST ≤ 2 times the upper limit of normal, serum total bilirubin ≤ 1.5 times normal Upper limit, serum creatinine ≥ 1.5 times normal upper limit, serum protein ≥ 30g / L; 6.At least one measurable lesion 7.There are no other serious diseases that conflict with this program, and the cardiopulmonary function is normal; 8.Women of childbearing age must have a negative urine or blood pregnancy test, and male patients should be contraceptive during medication; 9.There is no other antitumor treatment, but bisphosphonate for anti-bone metastasis treatment and other symptomatic treatment can be applied.

10.Can understand the situation of this study and sign the informed consent voluntarily

Exclusion Criteria:

1. rejecting providing blood preparation;
2. allergic to drug in this study or with hemophagocytic syndrome;
3. rejecting adopting reliable contraceptive method in pregnancy or lactation period;
4. uncontrolled internal medicine disease(including uncontrolled diabetes,severe incompetence cardiac,lung,liver and pancreas）；
5. with severe infection;
6. with primary or secondary central nervous system tumor invasion;
7. with Chemotherap or radiotherapy contraindication;
8. ever suffered with malignant tumor;
9. Human immunodeficiency virus (HIV)-positive patients
10. Drug abuse or long-term alcohol abuse that affects the evaluation of test results;
11. Have peripheral nervous system disorder or mental disorder;
12. Those who have no legal capacity or whose research is affected by medical or ethical reasons;

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months

SECONDARY OUTCOMES:
Time To Response (TTR) | Up to 3 months
Duration of Response (DOR) | Up to 2 years
Progression Free Survival (PFS) Progression Free Survival | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Professor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China